CLINICAL TRIAL: NCT01828905
Title: A Prospective, Multicenter, Randomized Study Investigating the Use of CERAMENT™|BONE VOID FILLER as Bone Graft Substitute in Tibia Plateau Fractures
Brief Title: Cerament Treatment of Fracture Defects
Acronym: CERTiFy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Univ.-Prof. Pol M. Rommens, Head of Department of Trauma Surgery, Director of the Center for Musculoskeletal Surgery, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S041/2012
Record Dates: First submitted 2013-04-04; First posted 2013-04-11 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: AO 41-B2 and AO 41-B3 Tibia Fractures
Keywords: tibia fracture; bone graft; iliac crest; bone graft substitute; Cerament; void filler; quality of life; pain; costs of care
MeSH Terms: conditions — Tibial Fractures; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cerament (Experimental): CERAMENT™|BONE VOID FILLER as bone graft substitute
  Interventions: Device: CERAMENT™|BONE VOID FILLER
- Bone graft (Active Comparator): Autologous cancellous bone graft (iliac crest)
  Interventions: Procedure: Autologous cancellous bone graft

INTERVENTIONS:
Device: CERAMENT™|BONE VOID FILLER — ceramic bone void filler
  Arms: Cerament
Procedure: Autologous cancellous bone graft — autologous cancellous bone graft
  Arms: Bone graft

SUMMARY:
The aim of the study is to compare fracture healing, quality of life, pain, and cost of care of the use of CERAMENT™|BONE VOID FILLER as bone graft substitute to the use of autologous cancellous bone graft (iliac crest) in the treatment of patients with tibia fractures treated by internal fixation and void reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* patients with traumatic, closed, depression fracture of the proximal tibia (limited to AO type B2 & B3)
* solitary trauma
* candidate for bone grafting
* patients between the age of 18 and 65 years
* written informed consent obtained before any study-related activities
* patients with communicative ability to understand the procedure and participate in the study and comply with the follow up program

Exclusion Criteria:

* patients with multiple injuries
* polytrauma patients
* compartment syndrome
* previous iliac crest bone graft harvesting
* local infection at the site of implantation
* chronic pain disease
* malignancy
* rheumatoid arthritis
* chronic cortisone intake
* X-ray diagnostics not available, fracture cannot be classified
* clinically significant or unstable medical or surgical condition that may preclude safe and complete study participation
* a pre-existing calcium metabolism disorder (e.g. hypercalcemia)
* known hyperthyroidism or autonomous thyroid adenoma
* history of serious reaction to iodine based radio contrast agents
* women who are pregnant or breastfeeding
* irreversible coagulopathy or bleeding disorder
* history of physical or psychological condition that contraindicates the use of an investigational device or render the patient at high risk from treatment complications
* history of hypersensitivity to the investigational device or any of its ingredients
* participation in other clinical trials during the present clinical trial or within the last 1 month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2013-04; Primary Completion 2017-12-24 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
SF-12 Physical Component Summary (PCS) at week 26 | 26 weeks
Global pain VAS score at week 26 | 26 weeks

SECONDARY OUTCOMES:
Utilisation of costs of care related resources | 26 weeks
SF-12 PCS and MCS at visit 4 | 1 week
Bone healing | 1, 6, 12 and 26 weeks
  Evaluated by X-ray
SF-12 PCS and MCS at visit 5 | 6 weeks
SF-12 PCS and MCS at visit 6 | 12 weeks
SF-12 PCS and MCS at visit 7 | 26 weeks

OTHER OUTCOMES:
Occurence of adverse events, device complaints and device-related incidents | 26 weeks
  Frequencies of subjects experiencing at least one adverse event (AE) will be displayed by body system and preferred term according to MedDRA terminology. Detailed information collected for each AE will include: a description of the event, duration, whether the AE was serious, intensity, relationship to trial device, action taken, clinical outcome. Summary tables will present the number of subjects observed with AEs and corresponding percentages.
  Number of device complaints and device-related incidents (AE related to the trial device) respectively as well as the frequencies of occurences of these events in both groups will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Pol M. Rommens, Univ.-Prof., MD, Principal Investigator — Department of Orthopaedics and Traumatology, Johannes Gutenberg University Mainz
Locations (16):
- Germany (16):
  - Clinic and Polyclinic for Trauma Surgery, Technical University München (Klinikum rechts der Isar), München, Bavaria
  - Clinic of Orthopaedics and Trauma Surgery, University Clinics of Freiburg, Freiburg im Breisgau, Geogr. Baden-Wuerttemberg
  - Clinic of Orthopaedics and Trauma Surgery, Hochtaunus-Kliniken gGmbH, Bad Homburg, Hesse
  - Clinic of Trauma, Hand and Reconstructive Surgery, University Clinics of Frankfurt, Frankfurt am Main, Hesse
  - Clinic of Orthopaedics and Trauma Surgery, Clinics of Fulda, Fulda, Hesse
  - Clinic of Trauma, Hand and Reconstructive Surgery, Healthcare Centre of Rüsselsheim (Gesundheits- und Pflegezentrum, GPR), Rüsselsheim am Main, Hesse
  - Clinic of Trauma, Hand and Reconstructive Surgery, University Clinics RWTH, Aachen, Northrhine-Westfalia
  - Clinic of Orthopaedics and Trauma Surgery, University Clinics of Cologne, Cologne, Northrhine-Westfalia
  - Clinic of Orthopaedics and Trauma Surgery, Occupational Accident Clinic (Berufsgenossenschaftliche Unfallklinik), Duisburg, Northrhine-Westfalia
  - Clinic of Trauma and Hand Surgery, University Clinics Düsseldorf, Düsseldorf, Northrhine-Westfalia
  - Clinic of Trauma, Hand and Reconstructive Surgery, Münster, Northrhine-Westfalia
  - Centre for Trauma Surgery and Orthopaedics, Stiftungsklinikum Mittelrhein, Koblenz, Rhineland-Palatinate
  - Clinic of Trauma Surgery and Orthopaedics, Occupational Accident Clinic (Berufsgenossenschaftliche Unfallklinik), Ludwigshafen am Rhein, Rhineland-Palatinate
  - Centre for Trauma surgery, Orthopaedics and Hand Surgery, Clinics of Worms, Worms, Rhineland-Palatinate
  - Department of Orthopaedics and Traumatology, Johannes Gutenberg University Mainz, Mainz, Rhineland-Palatine
  - Clinics of Musculoskeletal Surgery and Laboratory for Biomechanics, University of Schleswig-Holstein, Campus of Lübeck, Lübeck, Schleswig-Holstein

REFERENCES:
- [Background] Nusselt T, Hofmann A, Wachtlin D, Gorbulev S, Rommens PM. CERAMENT treatment of fracture defects (CERTiFy): protocol for a prospective, multicenter, randomized study investigating the use of CERAMENT BONE VOID FILLER in tibial plateau fractures. Trials. 2014 Mar 8;15:75. doi: 10.1186/1745-6215-15-75. PMID 24606670